CLINICAL TRIAL: NCT04686097
Title: Percutaneous Electrocoagulation Versus Sclerosing Foam for Patients With Incompetent Perforating Veins : A Multi-center Prospective Randomized Controlled Trial
Brief Title: Percutaneous Electrocoagulation Versus Sclerosing Foam for Patients With Incompetent Perforating Veins
Acronym: PESIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Shanghai Zhongshan Hospital (Other); Yantai Yuhuangding Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenjie Liu, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZhejiangU-003
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Incompetent Perforating Veins
Keywords: Perforating veins; Venous disease; Venous ulcer; Sclerotherapy; Electrocoagulationt
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (electrocoagulation) (Experimental): Participants in the experimental group will receive ultrasound-guided puncture of coagulation incompetent perforator veins.
  Interventions: Procedure: treatment: puncture of coagulation
- control group (sclerotherapy) (Active Comparator): Participants in the control group will receive an ultrasound-guided sclerosing agent injected.
  Interventions: Procedure: treatment: sclerosing agent injected

INTERVENTIONS:
Procedure: treatment: puncture of coagulation — ultrasound-guided puncture of coagulation
  Arms: experimental group (electrocoagulation)
Procedure: treatment: sclerosing agent injected — ultrasound-guided sclerosing agent injected
  Arms: control group (sclerotherapy)

SUMMARY:
This study aimed to compare the efficacy of punctured electrocoagulation and sclerotherapy in the treatment of incompetent perforator veins.

DETAILED DESCRIPTION:
Background: Incompetent perforating vein (IPV) is one of the important causes of persistent venous ulcers of lower extremities and recurrence after operation of varices which is a hot button issue worth discussing in clinical practice. Minimally invasive surgery has become the trend of IPVs' treatment. Currently, sclerotherapy can be performed to treat incompetent perforating veins, which showed a 90% occlusion rate after three or fewer sessions, the recurrence was present nearly 1/3 of cases. While electrocoagulation has a reliable effect on the closure of incompetent perforating veins and simplify treatment. No comparative studies of different PAPS modalities are currently available. Therefore, this study aimed to compare the efficacy of punctured electrocoagulation and sclerotherapy in the treatment of incompetent perforating veins. Methods:This study is a multicenter, randomized controlled trial. We will recruit 84 patients with IPVs from five hospitals. Moreover, these patients will be randomized to either the experimental group (electrocoagulation) or the control group (sclerotherapy). The primary outcome is incompetent perforating veins occlusion rate in the 12th month. Secondary outcomes are quality of life scale survey results (CEAP classification, VCSS score, CIVIQ-14 score), skin ulcer recurrence rate, deep venous Thrombosis, hemorrhage, all-cause mortality, and other vascular events and serious complications.Discussion:This study will provide reliable, evidence-based clinical evidence for the efficacy of electrocoagulation therapy for incompetent perforating veins.

ELIGIBILITY:
Inclusion Criteria:

(1) outward flow of less than 500 ms duration, with a diameter of >3.5 mm; (2) According to the CEAP classification method specified by the International Venous Federation, patients with C4b~C6 grades are included.

Exclusion Criteria:

(1)age < 18 years or age > 80 years; (2)with malignant tumors and life expectancy < 1 year; (3)with past or current history of deep vein thrombosis and/or pulmonary embolism in the lower extremities; (4)with congenital venous malformations (K-T syndrome, arteriovenous fistula and etc.; (5)inability to walk, long-term braking, restrictive bed rest; severe ischemia of lower extremities or diagnosed severity of peripheral artery occlusive disease; (6)according to the researcher's judgment, it is not suitable for foam hardener and puncture coagulation treatment; (7)allergic to the drugs and equipment materials involved in the research; (8)with inferior vena cava and/or iliac vein stenosis or occlusion; (9)with autoimmune disease, receiving chemotherapy, hormone therapy or immunomodulatory treatment; (10)other underlying severe diseases; women who are pregnant, breastfeeding or have pregnancy plans during the study period; (11)the patient cannot cooperate to complete the inspection and follow-up required by the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
IPVs occlusion rate in the 12th month. | 12 months after operation
  IPVs occlusion rate is defined as DS > 50% for each modality with no procedure no procedure performed on the treated segment

SECONDARY OUTCOMES:
Quality of life scale survey results | 1-month,6-month,12-month
  quality of life scale survey results (CEAP classification, VCSS score, CIVIQ-14 score).Quality of life will be assessed by MOS item short-form health survey scale (SF-36). SF-36 includes eight subscales: physical functioning (PF, 10 items), role limitations due to physical health problems (RL-P, 4 items), bodily pain (BP, 2 items), general health (GH, 5 items), vitality (V, 4 items), social functioning (SF, 2 items), role limitations due to emotional problems (RL-E, 3 items) and mental health (MH, 5 items). The vitality sub-score assesses energy and fatigue, and ranges from 0 (worst) - 100 (best).
Skin ulcer recurrence rate | 1-month,6-month,12-month
  Skin ulcer recurrence
Proportion of participants with deep venous Thrombosis | 1-month,6-month,12-month
  deep venous Thrombosis
Proportion of participants with hemorrhage | 1-month,6-month,12-month
  Including hemorrhagic stroke, gastrointestinal bleeding, hematuria, mucocutaneous hemorrhage and other visceral bleeding
All-cause mortality and other vascular events and serious complications. | 1-month,6-month,12-month
  Percentage of participants with all deaths

CONTACTS AND LOCATIONS:
Overall Officials: Zhen jie Liu, MD,PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (5):
- China (5):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang

REFERENCES:
- [Background] Cooper DG, Hillman-Cooper CS, Barker SG, Hollingsworth SJ. Primary varicose veins: the sapheno-femoral junction, distribution of varicosities and patterns of incompetence. Eur J Vasc Endovasc Surg. 2003 Jan;25(1):53-9. doi: 10.1053/ejvs.2002.1782. PMID 12525812
- [Background] Sakurai T, Matsushita M, Nishikimi N, Nimura Y. Hemodynamic assessment of femoropopliteal venous reflux in patients with primary varicose veins. J Vasc Surg. 1997 Aug;26(2):260-4. doi: 10.1016/s0741-5214(97)70187-3. PMID 9279313
- [Background] Guex JJ. Ultrasound guided sclerotherapy (USGS) for perforating veins (PV). Hawaii Med J. 2000 Jun;59(6):261-2. No abstract available. PMID 10916243
- [Background] Masuda EM, Kessler DM, Lurie F, Puggioni A, Kistner RL, Eklof B. The effect of ultrasound-guided sclerotherapy of incompetent perforator veins on venous clinical severity and disability scores. J Vasc Surg. 2006 Mar;43(3):551-6; discussion 556-7. doi: 10.1016/j.jvs.2005.11.038. PMID 16520171
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Hager ES, Washington C, Steinmetz A, Wu T, Singh M, Dillavou E. Factors that influence perforator vein closure rates using radiofrequency ablation, laser ablation, or foam sclerotherapy. J Vasc Surg Venous Lymphat Disord. 2016 Jan;4(1):51-6. doi: 10.1016/j.jvsv.2015.08.004. PMID 26946896